CLINICAL TRIAL: NCT03860688
Title: Investigating the Plasma Lipoprotein Response to a Single Subcutaneous Injection of Analogue Glucagon-like Peptide-2 and Oral Glucose in Humans
Brief Title: Effects of Oral Glucose and Teduglutide on Plasma Lipoproteins
Acronym: TED+GLC plasma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TED+GLC plasma 18-6296
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Hyperlipidemias
Keywords: Intestinal lipoprotein; Gut peptide; Chylomicrons; Glucose
MeSH Terms: conditions — Hyperlipidemias | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: On visit 2, participants will receive teduglutide and glucose 5 hours after a liquid meal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teduglutide + glucose (Experimental): Teduglutide, up to 0.05mg/kg, subcutaneous, single dose Glucose, 25g, oral, single dose
  Interventions: Drug: TED + glucose

INTERVENTIONS:
Drug: TED + glucose — Teduglutide, up to 0.05mg/kg, subcutaneous, single dose Glucose, 25g, oral, single dose

SUMMARY:
Some of the fat (triglyceride) from the food humans eat gets stored in the bowel. This triglyceride can then be released into the blood when another meal is consumed or in response to hormones. How the gut hormone glucagon-like peptide-2 (GLP-2) and glucose release the triglyceride from the gut is not known. The research team in this study is interested in finding out how teduglutide (a degradation resistant form of GLP-2) ang glucose, given together, release stored triglyceride from the gut by evaluating how blood lipoproteins respond to teduglutide in healthy individuals.

DETAILED DESCRIPTION:
The lipoprotein response will be performed in 15 healthy individuals recruited by newspaper advertisements. A member of the study team will explain the study in detail on visit 1, and if the individual is interested in participating, informed consent will be obtained and preliminary screening will occur. On visit 2 participants will receive a high fat liquid meal after an overnight fast. Hourly blood samples will be taken for 5 hours, followed by a subcutaneous teduglutide injection and simultaneous glucose drink. Following the injection and drink, blood samples will be taken every 15 minutes for the first hour and every 30 minutes for the subsequent 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years.
* Body mass index 20 to 27 kg/m2

Exclusion Criteria:

1. Patients with active inflammatory bowel disease
2. Patients with pre-existing Celiac disease, exocrine pancreatic insufficiency or small bowel malabsorption
3. Patients with active bowel malignancy
4. Patients with diabetes mellitus or known/ suspected motility disorders of the gut
5. Patients with decompensated liver disease
6. Patients on ezetimibe or bile acid sequestrants
7. Patients who are pregnant or breastfeeding.
8. Patients with renal disease.
9. Patients on benzodiazepine.
10. Unstable cardiac or respiratory disease
11. Any changes to medication in the preceding month
12. Patients with hypersensitive to Revestive or any ingredient, active or a history of the drug within the last 5 years
13. Patients with GI malignancy (GI tract, hepatobiliary, pancreatic)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Lipoprotein response to teduglutide and glucose | 8 hours
  To quantify the plasma lipoprotein response to teduglutide (GLP-2 analogue) injection and oral glucose in healthy individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No